CLINICAL TRIAL: NCT00151346
Title: Combined Spinal-Epidural Versus Traditional Labor Epidural: A Randomized, Controlled Trial Comparing Maternal and Fetal Effects
Brief Title: Combined Spinal-Epidural Versus Traditional Labor Epidural
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: New York Presbyterian Hospital (Other)
Responsible Party: Daniel W. Skupski, M.D., Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0306006204 (0603-889)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2008-03

CONDITIONS: Labour Pain
Keywords: Epidural; Labour pain; Pregnant women; Epidural anesthesia; Labour, Obstetric; labor pain; labor, obstetric; labor analgesia
MeSH Terms: conditions — Labor Pain | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CSE (Active Comparator): Subjects assigned to this group will receive "combined spinal-epidural" (CSE) to relieve pain during labor. For CSE, subjects receive a small amount of a local anesthetic and a small amount of a narcotic pain killer directly into the spinal canal (a smaller amount than is given for traditional epidural), followed by a small amount of both of these medications that is continuously infused into the epidural space through a catheter that is left in place. CSE is not experimental.
  Interventions: Drug: Bupivacaine and Fentanyl (for CSE)
- Traditional Epidural (Active Comparator): Subjects assigned to this group will receive "traditional epidural" to relieve pain during labor. For the traditional epidural, subjects receive a small amount of a local anesthetic and a small amount of a narcotic pain killer into the epidural space, followed by a small amount of both of these medications that is continuously infused into the epidural space through a catheter that is left in place. The traditional epidural is not experimental.
  Interventions: Drug: Bupivacaine and Fentanyl (for traditional epidural)

INTERVENTIONS:
Drug: Bupivacaine and Fentanyl (for CSE) — Bupivacaine 0.25% x 1 cc + Fentanyl 20 mcg, followed by infusion of Bupivacaine 0.0625% with Fentanyl 2 mcg/mL at 12 cc/hr
  Other Names: combined spinal-epidural; labor analgesia
  Arms: CSE
Drug: Bupivacaine and Fentanyl (for traditional epidural) — Bupivacaine 0.0625% with Fentanyl 2 mcg/mL x 15 cc, followed by infusion of Bupivacaine 0.0625% with Fentanyl 2 mcg/mL at 12 cc/hr
  Other Names: traditional epidural; labor analgesia
  Arms: Traditional Epidural

SUMMARY:
The purpose of this study to compare the use of spinal-epidural versus traditional labor epidural on maternal and fetal effects. The hope is to determine the safest and most effective epidural method of relieving pain during labor.

DETAILED DESCRIPTION:
Combined spinal-epidural anesthesia (CSE) was developed to allow excellent pain control for the pregnant woman who arrives in advanced labor and does not have much time for the anesthetic to have its effect. This has been extended recently to women in all stages of labor because of its rapid and excellent control of pain. Recent case series comparing CSE with traditional epidural have shown a slight difference in the rate of hypotension and fetal bradycardia, with the CSE technique having a higher rate of both of these side effects. This study will compare the two techniques in a prospective, randomized method.

The aim is to compare the maternal and fetal effects of two neuraxial block techniques for pain control during labor, to document blood pressure changes in upper and lower extremities pre- and post- block placement, and to document side effects (e.g. pruritus) and patient satisfaction with both techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read, understand and voluntarily sign the approved informed consent form (ICF) prior to any study- specific procedure;
* Must be between 18 to 50 years of age.
* Must be carrying a singleton fetus at term.
* Must have less than a body mass index of 40.
* Must be in labor, or is having a medical induction of labor.

Exclusion Criteria:

* Patient who has chronic renal disease, pre-existing hypertension, or pre-eclampsia.
* Patient who is undergoing an elective cesarean delivery
* Patient who has a presence of non-reassuring fetal status
* Patient who has an abnormal or non-reassuring fetal heart rate (FHR) pattern

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2003-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Adverse fetal effects: fetal bradycardia and abnormal fetal heart rate patterns | during the 60 minutes after placement of analgesia

SECONDARY OUTCOMES:
Average change in systolic blood pressure | during the 60 minutes after placement of analgesia
Average change in mean blood pressure | during the 60 minutes after placement of analgesia
Blood pressure differences between the upper and lower extremities | during the 60 minutes after placement of analgesia
Efficacy of analgesia as rated by the visual analog pain scale | during the 60 minutes after analgesic placement
Pruritus | through the first day following placement of analgesia
Incidence of hypotension | during the 60 minutes after placement of analgesia
Patient satisfaction | first day following placement of analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W. Skupski, M.D., Principal Investigator — Obstetrics & Gynecology; Weill Medical College of Cornell - New York Presbyterian Hospital; Klaus Kjaer-Pedersen, M.D., Principal Investigator — Anesthesiology; Weill Medical College of Cornell - New York Presbyterian Hospital
Locations (1):
- New York-Presbyterian Hospital; Weill Medical College of Cornell, New York, New York, United States